CLINICAL TRIAL: NCT05744388
Title: Efficacy of Lubricating the Under Surface of Glidescope Blade Stylet Shape Modification to Facilitate Endotracheal Intubation for Suspected Difficult Intubation; A Prospective Randomized Controlled Trial
Brief Title: Modification of the Stylet Shape of the Glidescope for Facilitating Difficult Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sabah Nageeb, Lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Glidescope
Record Dates: First submitted 2023-02-03; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Difficult Intubation
Keywords: difficult intubation; blade lubrication; stylet shape

STUDY DESIGN:
Intervention Model Description: Randomized prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stylet shape modification group (Active Comparator): Endotracheal tube diameter size 7.5 mm and disposable rigid blade size 3 for the female patients and ETT diameter size 8.00 mm and disposable rigid blade size 4 for the male patients will be prepared. The under surface of the blade will be lubricated by soluble jelly, taking care not to touch the camera source of light.
  The stylet will be more obtuse angle than the standard shape. The stylet will be lubricated also before being fitted inside the endotracheal tube. The blade will be introduced inside the mouth midline, the tube will be held from the upper third and introduced in the midline also sliding over the blade and introduced inside the glottis. Once the tip of the tube introduced inside the glottis, the stylet will be removed and the tube will be advanced more inside the trachea. The equality of air entry will be assessed by the stethoscope and the tube will by fixed by adhesive tape after inflating the cuff.
  Interventions: Device: Gliderite® shape modification
- Standard shape of the stylet group (No Intervention): The second group will be a control group, they will be handled by the standard shape of the stylet and the blade without lubrication.

INTERVENTIONS:
Device: Gliderite® shape modification — The stylet will be more obtuse angle than the standard shape. The stylet will be lubricated also before being fitted inside the endotracheal tube. The blade will be introduced inside the mouth midline, the tube will be held from the upper third and introduced in the midline also sliding over the blade and introduced inside the glottis.
  Other Names: Lubrication of the disposable blade by a jelly substance
  Arms: Stylet shape modification group

SUMMARY:
The undersurface of the disposable blade of the Glidescope will be lubricated by a jelly substance to facilitate its entrance to the mouth without trauma to the soft tissues. In addition the stylet ( Gliderite) shape will be modified to be an obtuse angle. This technique modification will be applied for obese patients with suspected difficult intubation criteria who are scheduled for bariatric surgeries.

DETAILED DESCRIPTION:
Endotracheal tube diameter size 7.5 mm and disposable rigid blade size 3 for the female patients and ETT diameter size 8.00 mm and disposable rigid blade size 4 for the male patients will be prepared. The under surface of the blade will be lubricated by soluble jelly, taking care not to touch the camera source of light.

The stylet will be more obtuse angle than the standard shape. The stylet will be lubricated also before being fitted inside the endotracheal tube. The blade will be introduced inside the mouth midline, the tube will be held from the upper third and introduced in the midline also sliding over the blade and introduced inside the glottis. Once the tip of the tube introduced inside the glottis, the stylet will be removed and the tube will be advanced more inside the trachea. The equality of air entry will be assessed by the stethoscope and the tube will by fixed by adhesive tape after inflating the cuff.

If during intubation the used technique failed to introduce the tube, we will do ETT rotation inside the mouth or upward stylet angulation outside the mouth then will be reintroduced again. If Glidescope failed to intubate, we will use intubating LMA to intubate the patients. If all trials failed to intubate the patients. Sugamadex 16 mg/Kg will be injected to awaken the patients. After intubation the large gastric tube will be introduced in the esophagus under vision by the Glidescope help also.

Group 2:

The second group will be a control group, they will be handled by the standard shape of the stylet and the blade without lubrication.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II or III
* BMI more than 35
* Patients presenting with at least one predictor for a difficult airway.
* The airway difficulty is at least score 3 as an indicator of difficulty.

Exclusion Criteria:

* Patients who may need rapid sequence induction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Intubation time in seconds | intraoperative time
  the intubation time will be calculated in seconds from the video screen of the Glidescope watch

SECONDARY OUTCOMES:
Number of trials of endotracheal intubation | intraoperative time
  the intubation time will be recorded
mucosal damage during the intubation | intraoperative time
  The blade under surface will be observed for blood spots. And the oral cavity will be viewed for mucosal damage or obscured view.

CONTACTS AND LOCATIONS:
Overall Officials: Sabah Ayoub, MD, Principal Investigator — Ain Shams University

REFERENCES:
- See also: 5. Ryo Wakabayashi1*, Yuki Shiko2 , Tomofumi Kodaira1 , Yuko Shiroshita1 , Hitomi Otsuka1 , Kosuke Baba1 & Norimasa Hishinuma Efcacy of stylet angulation at the holding position during tracheal intubation with a videolaryngoscope: a randomized controlled — https://doi.org/10.1038/s41598-021-00115-x